CLINICAL TRIAL: NCT03043755
Title: Observational Study to Evaluated Efficacy of Parasternal and PECS Blocks Association in Breast Surgery
Brief Title: PECS and Parasternal Block for Breast Surgery
Acronym: PARAST
Status: Completed | Type: Observational
Sponsor: Istituti Ospitalieri di Cremona (Other)
Responsible Party: Principal Investigator, Erika Basso Ricci, Anesthetist, Istituti Ospitalieri di Cremona
Other Study IDs: ANECR_01_17
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Quadrantectomy; Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Propose to evaluate efficacy of association between US guide parasternal block and pectorals nerves block (PECS) as anesthetic option for breast surgery (medial quadrantectomy and simple mastectomy).

All patients undergoing medial quadrantectomy and simple mastectomy in 6 months period will be observed.

All patients receive: US guide parasternal block at T4 and T6 space with 6ml of ropivacaine 0,75% and PECS type 2 block performed with 24ml of ropivacaine 0,75%.

During surgery patients receive light sedation with continuous infusion of propofol

Will be observed:

Additional local anesthetic infiltration from surgeon. Pain at rest and during movement quantified as Numerical Rating Scores (0-10) during the first 12 hours postoperatively.

Eventual side effects such as nausea/vomiting.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years;
* ASA score I - II - III;
* undergoing elective medial quadrantectomy breast surgery;
* undergoing elective mastectomy not reconstruction breast surgery;
* signed informed consent;

Exclusion Criteria:

* chronic therapy with opioids/ antidepressants;
* urgent/emergent surgery;
* postoperative transfer to the intensive care unit;
* known allergy to any drug medication;
* local skin infection;
* epilepsy;
* alcohol or drug abuse;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing breast surgery
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Local Anesthetic infiltration | intraoperatory period
  Quantify amount of local anesthetic infiltration from surgeon to get perfect anesthesia
Convention in general anesthesia | preoperative period
  Number of patients require general anestesia to proceed to surgery

SECONDARY OUTCOMES:
Pain | 12 hours postoperatively
  Rest and in mouvement pain as NRS scale
PONV | 12 hours postoperatively
  Postoperative nausea/vomiting incidence

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Cremona, Creom, Cremona, Italy

IPD SHARING:
Plan to Share IPD: No